CLINICAL TRIAL: NCT03544086
Title: Clinical Evaluation of a Wearable Sleep Diagnosis Technology
Status: Completed | Type: Observational
Sponsor: Acurable Ltd. (Industry)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 225818; 225818 (Other: IRAS)
Record Dates: First submitted 2018-05-22; First posted 2018-06-01 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- test group: First group is the first 10 patients
- study group: following 150 patients

SUMMARY:
The primary endpoint is to evaluate the sensitivities and specificities for diagnosis of sleep apnoea of a wearable sleep diagnosis technology vs. existing gold standard.

DETAILED DESCRIPTION:
The clinical investigation will be performed at the Royal Free London Hospital. Physiological signals will be pseudo-anonymized and only viewed by the research team.

The Study will involve patients who will have been referred for diagnosis of sleep apnoea, will aim to determine AcuPebble's positive and negative predictive ratios, sensitivities as specificities. Likelihood ratios for diagnosis of sleep apnoea. Clinical experts will determine patients' diagnostic information using the current diagnostic standards. AcuPebble will also generate diagnostic results independently and automatically. Both set of results will be subsequently compared and the relevant performance metrics listed above will be determined.

Consecutive patients referred for sleep study will be recruited to the study. Patients that are willing to participate will be consented on the day of their sleep study and sent home with both - the Trusts usual multichannel polygraphy and the Acupebble.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been referred to a sleep clinic due to suspicion of sleep apnoea.

Exclusion Criteria:

* Age under 18 or over 70 years.
* Subjects who are not fluent in English, or who have special communication needs.
* Known allergy to the adhesive dressing.
* Subjects with physical or mental impairments who would not be able to use the new technology on their own.
* Subjects with very loose/saggy skin in the neck area which would unavoidably result on - AcuPebble swinging if moving the neck.
* Subjects with pacemakers.
* exclude patients who have any type of implanted electronic devices (these include patients in ICDs and left ventricular assist devices and loop recorders).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been referred to a sleep clinic due to suspicion of sleep apnoea, consecutive 160 patients coming to the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Sensitivities and Specificities for diagnosis of sleep apnoea studies | 6 months
  Sensitivities and Specificities for diagnosis of sleep apnoea studies

CONTACTS AND LOCATIONS:
Overall Officials: Dr Swapna Mandal, BSc MBBS MRCP SCE, PhD, Principal Investigator — Royal Free NHS Hospital
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Devani N, Pramono RXA, Imtiaz SA, Bowyer S, Rodriguez-Villegas E, Mandal S. Accuracy and usability of AcuPebble SA100 for automated diagnosis of obstructive sleep apnoea in the home environment setting: an evaluation study. BMJ Open. 2021 Dec 21;11(12):e046803. doi: 10.1136/bmjopen-2020-046803. PMID 34933855